CLINICAL TRIAL: NCT06010381
Title: Muscle Energy Technique Versus Maitland Mobilization on Shoulder Pain and Disability After Neck Dissection Surgeries.
Brief Title: Muscle Energy Technique Versus Maitland Mobilization on Shoulder Pain and Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003370
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Neck Cancer; Mobility Limitation; Pain Syndrome; Shoulder Pain; Surgery
Keywords: Muscle energy technique; Maitland's mobilization; shoulder pain and disability; neck dissection surgeries
MeSH Terms: conditions — Head and Neck Neoplasms; Mobility Limitation; Somatoform Disorders; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Patients were subdivided into two groups, fifteen patients in each group. Group A received the muscle energy technique and group B received Maitland's mobilization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle energy technique (Active Comparator): This group includes 15 patients who received muscle energy technique post-surgery in addition to traditional shoulder exercise, 3 sessions/week for four weeks.
  Interventions: Other: Muscle energy technique; Other: Traditional shoulder exercise
- Maitland mobilization (Active Comparator): This group includes 15 patients who received mobilization in addition to traditional shoulder exercise, 3 sessions/week for four weeks.
  Interventions: Other: Maitland mobilization; Other: Traditional shoulder exercise

INTERVENTIONS:
Other: Muscle energy technique — It was applied on the shoulder flexion and the external rotation. An isometric contraction of the agonist muscle (the muscle which requires stretching) for 7 seconds with gentle muscle contraction to avoid the risk of increasing the muscle tone. This contraction started just short of the restrictive barrier. After that, the patient is asked to relax for 2-3 seconds and then the therapist stretches the contracted muscle in the opposite direction for 30 seconds. This is repeated three repetitions for each muscle.
  Arms: Muscle energy technique
Other: Maitland mobilization — At the start of each session, the physical therapist examined the patient's ROM in all directions to obtain information about the end-range position and the end feel of the glenohumeral joint. Start with rhythmic mid-range mobilization with the patient in a supine position. The therapist's hands are placed close to the glenohumeral joint, and the humerus is brought into a position of maximal flexion in the sagittal plane. After 10 to 15 repetitions of intensive mobilization techniques in this end-range position, the direction of mobilization will be altered by varying the plane of elevation or by varying the degree of rotation. When alternating the direction of mobilization, other movements such as gliding techniques and distraction in that joint position were (inferior gliding, anterior gliding, and posterior gliding).
  Arms: Maitland mobilization
Other: Traditional shoulder exercise — Traditional shoulder exercises in the form of shoulder range of motion exercises, stretching exercises and, scapular stabilization.

SUMMARY:
The purpose of this study was to investigate the effect of muscle energy technique versus Maitland's mobilization on shoulder pain and disability after neck dissection surgeries.

DETAILED DESCRIPTION:
Thirty patients with shoulder pain and limited ROM post-neck dissection surgeries participated in this study. Patients were subdivided into two groups, fifteen patients in each group. Group A received the muscle energy technique and group B received Maitland's mobilization.

Data obtained from both groups regarding the Visual Analogue Scale, it has a 100-mm-long horizontal line labeled ''no pain' (with or without related facial expressions) at one extreme and ''worst pain ever' at the other. Pain intensity is determined by the length of the line as measured from the left-hand side to the point marked, The Shoulder Pain and Disability Index, it has two subscales; The pain subscale includes five questions about pain intensity. The disability subscale includes eight questions about difficulty in different orders. Each question of both pain and disability subscale was scaled in numeric ratings ranging from 0 to 10. Each score was summed up and transformed into percentages. Finally, the average score between pain and disability subscale comprised the total SPADI scores ranging from 0 (the best) to 100 (the worst), and shoulder flexion, abduction, and external ROM were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 25-70 years.
* Male and female patients participated in the study.
* All patients had shoulder pain following different NDS
* All patients had no previous shoulder pain.
* All patients enrolled in the study had their informed consent.

Exclusion Criteria:

* Previous shoulder pain from any other causes.
* Pregnancy.
* Epileptics.
* Radiotherapy.
* Chemotherapy.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | Change from baseline at four weeks after the intervention
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiology and clinical research to measure the intensity or frequency of various symptoms. It has a 100-mm-long horizontal line labeled ''no pain' (with or without related facial expressions) at one extreme and ''worst pain ever' at the other. Pain intensity is determined by the length of the line as measured from the left-hand side to the point marked.
Shoulder Pain and Disability Index | Change from baseline at four weeks after the intervention
  It is a self-reported questionnaire consisting of 13 items divided in two parts: pain and disability sub-scale. The pain subscale includes five questions about pain intensity. The disability subscale includes eight questions about difficulty in different orders. Each question of both pain and disability subscale was scaled in numeric ratings ranging from 0 to 10. Each score was summed up and transformed into percentages. Finally, the average score between pain and disability subscale comprised the total SPADI scores ranging from 0 (the best) to 100 (the worst).
Shoulder active range of motion | Change from baseline at four weeks after the intervention
  Through using the universal goniometer to measure the shoulder flexion, abduction and, external rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA El Sayeh, PhD, Study Director — Lecturer at Faculty of Physical Therapy, Cairo University
Locations (1):
- Shaimaa Mohamed Ahmed El Sayeh, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No